CLINICAL TRIAL: NCT00358319
Title: Phase I/II Trial of Valproic Acid and Karenitecin for Metastatic Malignant Melanoma
Brief Title: Phase I/II Trial of Valproic Acid and Karenitecin for Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left Moffitt
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: BioNumerik Pharmaceuticals, Inc. (Industry)
Responsible Party: Adil Daud, M.D., UCSF (formerly with H. Lee Moffitt Cancer Center and Research Institute)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-13991
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2011-02

CONDITIONS: Malignant Melanoma
Keywords: Valproic Acid (VPA); Karenitecin; Malignant Melanoma; Histone deacetylases (HDAC)inhibitors; Topoisomerase I inhibitor; metastatic
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — cositecan; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phase I (Experimental): Dose escalation phase
  Interventions: Drug: Karenitecin; Drug: Valproic Acid
- Phase II (Experimental): All patients enrolled in the Phase II will be treated with Valproic Acid (VPA) and Karenitecin using the dosing schedule determined to be the Maximum Tolerated Dose (MTD) in Phase I.
  Interventions: Drug: Karenitecin; Drug: Valproic Acid

INTERVENTIONS:
Drug: Karenitecin
Drug: Valproic Acid
  Other Names: VPA

SUMMARY:
This is a Phase I study looking at the combination of Valproic Acid (VPA) and Karenitecin to treat patients with metastatic malignant melanoma. We will find the dose-limiting toxicity (DLT) and the highest dose (maximum tolerated dose) of this combination treatment that has acceptable side effects and recommend a Phase II dose level.

There will be seven escalating doses of Valproic acid and one dose escalation step of Karenitecin. Each patient shall receive one cycle of Karenitecin alone (cycle 1 days 1 - 5) followed by the same dose of Karenitecin given in combination with VPA (cycle 2 days 1-7). Patients will receive oral VPA in divided doses for 5 days and Karenitecin starting on the 3rd day every 3 weeks (a treatment cycle).

Treatment will continue until progression of disease or an unacceptable level of toxicity. After 2 cycles of treatment there will be the first efficacy evaluation or restaging of the disease. In the absence of disease progression and if there is continued safety and tolerability, treatment may continue.

DETAILED DESCRIPTION:
Treatment cycles are every 3 weeks and there are 17 study visits in all.

During Phase I subjects will receive one cycle of Karenitecin alone (cycle 1 days 1-5) and then combination therapy with VPA + Karenitecin (cycle 2 days 1-7)followed by oral VPA in divided doses for 5 days and Karenitecin starting the third day (days 3-7) every 3 weeks. After 2 cycles of treatment there will be the first efficacy evaluation or restaging of the disease.

Dose escalations will continue until unacceptable dose limiting toxicity (DLT) occurs, then dose escalation will be stopped and the previous dose level will be explored. In each dose level, participants will undergo pharmacokinetic (PK) sampling to determine blood levels. The melanoma skin lesions will also be biopsied to measure the effect of the combination therapy.

All patients enrolled in the Phase II will be treated with VPA and Karenitecin using the dosing schedule determined to be the MTD in Phase I. In the absence of disease progression and if there is continued safety and tolerability, treatment may continue in consecutive 3 week cycles.

ELIGIBILITY:
Inclusion Criteria:

Same for Phase I & II

* Cytologically/histologically-documented metastatic (stage IV) malignant melanoma
* Age greater than or equal to 18 years old
* ECOG performance status 0-2
* Subjects must be able to give informed consent and be able to follow the guidelines given in the study
* The subject has no major impairment of hematological function, as defined by the following laboratory parameters: WBC > 3.0x109/L; ANC > 1.5 x 109/L; Hgb > 9.0g/dL; PLT >100x109/L. Red blood cell transfusions and repeat evaluations for study entry are allowed
* All subjects of reproductive potential must use an effective method of contraception during the study and three months following termination of treatment (Not applicable to patients with bilateral oophorectomy and/or hysterectomy or to those patients who are postmenopausal.)
* Subjects with biopsiable disease are preferred but not mandatory; subjects with biopsiable disease will be encouraged to undergo biopsy.

Exclusion Criteria:

Phase I:

* Subjects must not have evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry.
* Subjects must have adequate renal and normal hepatic function (creatinine < 1.5 x upper limit of normal (ULN), bilirubin and SGOT (AST) < 1.5 X ULN) obtained within 4 weeks prior to registration.
* Pregnant women are excluded from the study because VPA is known to cause birth defects. Nursing mothers are excluded from this trial as effects on newborns and excretion of either drug in milk is unknown.
* Women of childbearing age must have a negative pregnancy test and be willing to use a highly effective method of contraception. Men who are sexually active must also be willing to use an accepted and effective method of contraception.
* Subjects with uncontrolled CNS metastasis or a history of seizures are excluded. Subjects with stable CNS metastasis (either surgically resected, treated with the gamma knife or stable for 3 months following whole brain radiotherapy are eligible)

Phase II:

* Subjects must not have evidence of significant active infection (e.g., pneumonia, cellulitis, wound abscess, etc.) at time of study entry.
* Subjects must have adequate renal and normal hepatic function (creatinine < 1.5 x upper limit of normal (ULN), bilirubin and SGOT (AST) < 1.5 X ULN) obtained within 4 weeks prior to registration.
* Pregnant women are excluded from the study because VPA is known to cause birth defects. Nursing mothers are excluded from this trial as effects on newborns and excretion of either drug in milk is unknown.
* Women of childbearing age must have a negative pregnancy test and be willing to use a highly effective method of contraception. Men who are sexually active must also be willing to use an accepted and effective method of contraception.
* Subjects with uncontrolled CNS metastasis or a history of seizures are excluded. Subjects with stable CNS metastasis (either surgically resected, treated with the gamma knife or stable for 3 months following whole brain radiotherapy are eligible)
* Subjects who have been previously treated with more than 2 prior chemotherapy regimens. Any previous immunotherapy regimens are allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-03; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety profile of Valproic Acid (VPA) and Karenitecin | Average of 6 months
Maximum tolerated dose (MTD) of Valproic Acid and Karenitecin | Average of 6 months
Response rate | Average of 6 months
Time to progression (TTP) | Average of 6 months
Overall survival (OS) | Average of 6 months

SECONDARY OUTCOMES:
Pharmacokinetic parameters of VPA and Karenitecin | Average of 6 months
Relationship between topo I expression, location and DNA strand breakage | Average of 6 months
Patient response to this drug combination | Average of 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Adil Daud, M.D., Principal Investigator — UCSF (formerly at H. Lee Moffitt Cancer Center & Research Institute)
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States